CLINICAL TRIAL: NCT01330420
Title: Outcomes and Cost-Effectiveness of a Behavioral Medicine Intervention With Depressed Patients in a Community Health Center Setting
Brief Title: Behavioral Medicine Intervention With Depressed Patients in a Community Health Center Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, John W. Denninger, MD, PhD, Director of Research at the Benson-Henry Institute for Mind Body Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007P001633; Center for Disease Control (Other Grant/Funding Number: 5R01DP000339)
Record Dates: First submitted 2011-03-11; First posted 2011-04-07 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Meditation; Cognitive Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Relaxation Response Resiliency Program for Depression (Experimental): The Relaxation Response Resiliency Program for Depression (3RP-D) is a low-cost, easily replicable, 6-session, 1.5 hour, mind body intervention.
  The 3RP-D was designed to promote resiliency by reducing the harmful effects of stress through the elicitation of the relaxation response, and through skill training to enhance positive attitudes and beliefs, nutrition, exercise, recuperative sleep, social support, and coping. Specific interventions include: cognitive behavioral therapy (CBT), enhancing social support (SS), cultivating positive attitudes and beliefs (CPE), and promoting Healthy Lifestyle Habits(HL). The 3RP-D program has been manualized for use by group facilitators and health center patients.
  Interventions: Behavioral: Relaxation Response Resiliency Program for Depression

INTERVENTIONS:
Behavioral: Relaxation Response Resiliency Program for Depression — The program combines lecture, skills training, symptom monitoring, and group sharing aimed at preparing patients to take active roles in managing their own health. Elements of the program include:
  * Elicitation of the relaxation response through techniques such as diaphragmatic breathing and mindfulness.
  * Examination and reversal of negative thought patterns.
  * Physical movement, including stretching and yoga.
  * Healthy eating and other positive lifestyle behaviors.
  * Goal setting.
  Other Names: Medical Symptom Reduction Program, Meditation, Mind Body techniques, Cognitive Psychology

SUMMARY:
The linkage between the Massachusetts General Hospital (MGH)-Community Health Associates and the MGH-Benson Henry Institute for Mind-Body Medicine began in order to address the concern of providing affordable, easily accessible, culturally appropriate behavioral medicine interventions for low income patients served by MGH Community Health Centers, as well as the desire to demonstrate the efficacy and economics of these interventions. Since depression was such a prevalent issue among health center patients, with a significant impact on health care service utilization, it was decided to focus on offering Mind/Body services to this population first.

DETAILED DESCRIPTION:
The application of behavioral medicine programs in community health settings is important to explore, as that application empowers the patient to apply self-care modalities that can be utilized in the long-term, for depression as well as for many other stress-related illnesses.

Behavioral and Mind/Body techniques, such as the Relaxation Response, have been reported to be useful therapeutically (often as an adjunct to medical treatment) in numerous conditions that are caused or exacerbated by stress including: mild to moderate depression/anxiety; anxiety; headache; back/neck pain; myocardial ischemia; premature ventricular contractions in stable ischemic heart disease or hypertension; osteoarthritis; stress symptoms; improved outcomes after cardiac and other surgery; pain relief and anxiety reduction in femoral arteriography and other invasive medical procedures; premenstrual syndrome; infertility; psychosomatic complaints; chronic pain; insomnia; musculoskeletal disorders; wound healing; rheumatoid arthritis; fibromyalgia and disease and treatment related symptoms of cancer. In our recent review of the literature, we suggest that the Relaxation Response may be an appropriate and relevant therapeutic state to counteract several stress-related disease processes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 21 years of age or older
* Diagnosis of depression
* Currently being treated for depression with medications and/or psychological counseling through one of the MGH-HealthCare Centers.
* Planning to continue using the health center as their main source of general medical services for the coming year.

Exclusion Criteria:

* History of bipolar disorder
* Active substance abuse
* History of psychosis
* Severe cognitive dysfunction (MMSE ≤ 24)
* Inability to speak English
* We will not exclude patients on the basis of their religious preferences or practices.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-09; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L. Fricchione, MD, Principal Investigator — Massachusetts General Hospital; Kathleen M. Miller, RN, Study Director — Massachusetts General Hospital; Herbert Benson, MD, Study Director — Massachusetts General Hospital; John W. Denninger, MD, PhD, Study Director — Massachusetts General Hospital
Locations (2):
- United States (2):
  - MGH Community Health Care Center, Charlestown, Massachusetts
  - MGH Community Health Care Centers, Revere, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were being treated for depression with medications or psychotherapy at the MGH-Revere or MGH-Charlestown Health Centers. Referrals came from health center primary care providers (PCP's), mental health providers, or directly from patients themselves through postcards in the waiting areas.
Pre-assignment Details: Licensed independent clinical social worker (LICSW) Group Facilitators administered intake evaluations with the referred patients to obtain basic demographic and clinical information, determine if they were appropriate for the group based on the inclusion and exclusion criteria, and review their goals for group participation.
Groups:
- Relaxation Response Resiliency Program for Depression: The Relaxation Response Resiliency Program for Depression (3RP-D) is a low-cost, easily replicable, 6-session mind body intervention that was derived from the Medical Symptom Reduction Program (MSRP), an earlier iteration of the BHI's current Relaxation Response Resiliency Program (3RP.)
  The cornerstone of the 3RP-D is elicitation of the relaxation response, and this approach is reinforced by additional resiliency-enhancing interventions including group Cognitive Behavioral Therapy (CBT), Positive Psychology and cultivation of Conscious Positive Expectation (CPE), Social Support (SS), and promotion of Healthy Lifestyle behaviors (HL).
Period: Overall Study
Arm/Group | Relaxation Response Resiliency Program for Depression
Started | 28
Completed | 24
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Relaxation Response Resiliency Program for Depression
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Depression Severity (CEDS-10)
Description: The Center for Epidemiologic Studies Depression Scale (CES-D 10) was used to assess depression severity pre-and post-intervention. This is the shorter 10-item, modified version of the 20-item CES-D. The total score is the sum of the 10 item weights, with the lowest possible score being 0 and the highest possible score being 30, and a higher score indicating more depressive symptoms. Developed from other well-validated depression scales, this instrument measures the experience of depressive symptoms over the past week. This instrument is shown to be better than the CES-D 20 in combining data from different ethnic and cultural groups, and is available in both English and Spanish. This scale has been reported to have good internal consistency and validity.
Time Frame: comparison pre program initiation and post program completion time points (6 weeks)
Population: 24 patients met completer status, defined as patients who attended all or part of the six sessions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Response Resiliency Program for Depression
Number analyzed (Participants) | 24
units on a scale
  CSE-D 10 Pre-Intervention | 18 (5.8)
  CSE-D 10 Post-Intervention | 12 (5.7)
Statistical Analysis 1: Comparison: Relaxation Response Resiliency Program for Depression; Due to the small sample size, the Wilcoxon signed-ranked test, a non-parametric statistical test, was used to detect outcome measure changes from pre-intervention to post-intervention; Test type: Superiority or Other; p < .001, Wilcoxon signed-ranked test

2. Primary Outcome: Health Status (SF-12)
Description: The SF-12 was used to assess health status. It is the shortened version of the well-validated SF-36, directed at monitoring overall physical and mental health outcomes. It is available in both English and Spanish. Scoring algorithms involve weighted-item responses, all 8 scales to use the same standardization for easy comparison. All scores range from 0-100 where higher scores indicated better QOL. The mean = 50 and the SD = 10.
Time Frame: comparison pre program initiation and post program completion time points (6 weeks)
Population: 24 patients met completer status, defined as patients who attended all or part of the six sessions. Not all 24 patients had complete pre-/post-intervention questionnaires sets. Therefore, patients may have missed some of the questionnaires, either pre- or post-intervention, and thus the number of patients analyzed maybe less than 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Response Resiliency Program for Depression
Number analyzed (Participants) | 23
units on a scale
  SF-12 General Health Pre-Intervention | 51 (24)
  SF-12 General Health Post-Intervention | 49 (28)
  SF-12 Physical Functioning Pre-Intervention | 58 (38)
  SF-12 Physical Functioning Post-Intervention | 58 (35)
  SF-12 Role Physical Pre-Intervention | 65 (44)
  SF-12 Role Physical Post-Intervention | 61 (43)
  SF-12 Role Emotional Pre-Intervention | 17 (39)
  SF-12 Role Emotional Post-Intervention | 39 (50)
  SF-12 Bodily Pain Pre-Intervention | 62 (34)
  SF-12 Bodily Pain Post-Intervention | 59 (37)
  SF-12 Mental Health Pre-Intervention | 34 (17)
  SF-12 Mental Health Post-Intervention | 50 (20)
  SF-12 Vitality Pre-Intervention | 30 (16)
  SF-12 Vitality Post-Intervention | 39 (24)
  SF-12 Social Functioning Pre-Intervention | 48 (29)
  SF-12 Social Functioning Post-Intervention | 59 (25)
Statistical Analysis 1: Comparison: Relaxation Response Resiliency Program for Depression; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .001, Wilcoxon signed-ranked test

3. Primary Outcome: Quality of Life (QOL-5)
Description: The QOL-5 is a short, global, and generic quality of life (QoL) questionnaire for clinical databases. The QOL-5 item tool is used to compare various population groups using generic factors common to people everywhere irrespective of age, sex, culture, and state of health. Scores on the QOL-5 ranges from 0 = lowest quality to 100 = highest quality.
Time Frame: comparison pre program initiation and post program completion time points (6 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Response Resiliency Program for Depression
Number analyzed (Participants) | 24
units on a scale
  QoL-5 Pre-Intervention | 56 (9.9)
  QoL-5 Post-Intervention | 62 (12)
Statistical Analysis 1: Comparison: Relaxation Response Resiliency Program for Depression; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .01, Wilcoxon signed-ranked test

4. Primary Outcome: Satisfaction With Care (PSQ-18)
Description: Patient Satisfaction Questionnaire Short Form (PSQ-18) takes approximately 3-4 minutes to complete, containing 18 items examining seven dimensions of satisfaction with medical care: general satisfaction (2 questions, Mean =3.58, SD =0.94), technical quality (3 questions, Mean = 3.68, SD = 0.76), interpersonal manner (2 questions, Mean = 4.09, SD = 0.69), communication (2 questions, Mean = 3.74, SD = 0.87), financial aspects (2 questions, Mean = 3.78, SD = 0.94), time spent with doctor (2 questions, Mean = 3.59, SD = 0.94), and accessibility and convenience (4 questions, Mean = 3.76, SD = 0.74). Responses to each item are given on a 5-point scale ranging from 1 - strongly agree to 5 - strong disagree, therefore higher scores correspond to less satisfaction. PSQ-18 subscale scores are substantially correlated with their full-scale counterparts and possess generally adequate internal consistency reliability.
Time Frame: comparison pre program initiation and post program completion time points (6 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Response Resiliency Program for Depression
Number analyzed (Participants) | 22
units on a scale
  PSQ-18 General Satisfaction Pre-Intervention | 3.9 (0.8)
  PSQ-18 General Satisfaction Post-Intervention | 3.8 (0.8)
  PSQ-18 Technical Quality Pre-Intervention | 4.0 (0.6)
  PSQ-18 Technical Quality Post-Intervention | 3.7 (0.6)
  PSQ-18 Interpersonal Manner Pre-Intervention | 4.3 (0.6)
  PSQ-18 Interpersonal Manner Post-Intervention | 4.1 (0.8)
  PSQ-18 Communication Pre-Intervention | 4.0 (0.7)
  PSQ-18 Communication Post-Intervention | 3.8 (0.8)
  PSQ-18 Financial Aspects Pre-Intervention | 3.8 (1.1)
  PSQ-18 Financial Aspects Post-Intervention | 3.8 (1.0)
  PSQ-18 Time Spent with Doctor Pre-Intervention | 3.9 (0.6)
  PSQ-18 Time Spent with Doctor Post-Intervention | 3.7 (0.9)
  PSQ-18 Accessibility & Convenience Pre-Inter. | 3.4 (0.9)
  PSQ-18 Accessibility & Convenience Post-Inter. | 3.3 (0.7)

5. Secondary Outcome: The Health Promoting Lifestyle Profile II (HPLP-II)
Description: The Health Promoting Lifestyle Profile II (HPLP-II) was used to assess health promoting behaviors. Based on the Health Promoting Model (Pender, 1982) this 52-item instrument measures self-initiated health behaviors that serve to maintain or enhance the level of self-actualization and wellness. Included are subscales for physical activity, spiritual growth, health responsibility, interpersonal relations, nutrition, and stress management. It is self-administered and uses a 4-point response format. Both English and Spanish versions are available.
  A score for overall health-promoting lifestyle is obtained by calculating a mean of the individual's responses to all 52 items; six subscale scores are obtained similarly by calculating a mean of the responses to subscale items. Scores range from 1 = Never to 4 = Routinely, with a higher score corresponding to a more health promoting lifestyle.
Time Frame: comparison pre program initiation and post program completion time points (6 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Response Resiliency Program for Depression
Number analyzed (Participants) | 23
units on a scale
  HPLP II - Spiritual Growth Pre-Intervention | 2.0 (0.5)
  HPLP II - Spiritual Growth Post-Intervention | 2.4 (0.7)
  HPLP II - Health Responsibility Pre-Intervention | 2.7 (0.6)
  HPLP II - Health Responsibility Post-Intervention | 2.7 (0.5)
  HPLP II - Physical Activity Pre-Intervention | 1.9 (0.7)
  HPLP II - Physical Activity Post-Intervention | 2.2 (0.8)
  HPLP II - Nutrition Pre-Intervention | 2.6 (0.6)
  HPLP II - Nutrition Post-Intervention | 2.5 (0.6)
  HPLP II - Interpersonal Relations Pre-Intervention | 2.7 (0.5)
  HPLP II - Interpersonal Relations Post-Inter. | 2.8 (0.5)
  HPLP II - Stress Management Pre-Intervention | 2.1 (0.5)
  HPLP II - Stress Management Post-Intervention | 2.5 (0.6)
Statistical Analysis 1: Comparison: Relaxation Response Resiliency Program for Depression; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .01, Wilcoxon signed-ranked test

ADVERSE EVENTS:
Arm/Group | Relaxation Response Resiliency Program for Depression
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

LIMITATIONS AND CAVEATS:
4/28 didn't complete both pre/post assessments & thus didn't contribute data for this study & were excluded. It's possible that the 24 completers had a higher degree of motivation & commitment, which enhanced the effectiveness of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No